CLINICAL TRIAL: NCT00687544
Title: Efficacy and Safety of PegIntron Plus Ribavirin for Treatment of Chronic Hepatitis C Infection in HIV-Infected Persons Not Previously Treated With Interferon
Brief Title: Efficacy and Safety of PegIntron Plus Ribavirin for Treatment of Chronic Hepatitis C in HIV-Infected Subjects (Study P04469)(TERMINATED)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04469
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic; Hepacivirus; HIV Infections
Keywords: HIV
MeSH Terms: conditions — Hepatitis C, Chronic; HIV Infections | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEG-IFN + RBV (Experimental): PEG-IFN + RBV therapy in previously untreated chronic HCV subjects coinfected with HIV
  Interventions: Biological: Peginterferon alfa-2b (SCH 054031); Drug: Ribavirin (SCH 018908)

INTERVENTIONS:
Biological: Peginterferon alfa-2b (SCH 054031) — Subjects will be given peginterferon alfa-2b (PEG-IFN) subcutaneously, at a dose of 1.5 ug/kg weekly. Treatment duration will be 48 weeks for subjects with Hepatitis C Virus (HCV) genotype 1 and 24 weeks for subjects with HCV genotype 2 or 3 and baseline Hepatitis C Virus-ribonucleic acid (HCV-RNA) below 800,000 IU/mL.
  Other Names: PegIntron
Drug: Ribavirin (SCH 018908) — Subjects will be given ribavirin 800 mg/day orally(PO) when body weight is <65 kg, 1000 mg/day when body weight is between 65 kg and 85 kg, and 1200 mg/day when body weight is >85 kg. Treatment duration will be 48 weeks for subjects with HCV genotype 1 and 24 weeks for subjects with HCV genotype 2 or 3 and baseline HCV-RNA below 800,000 IU/mL.
  Other Names: Rebetol

SUMMARY:
In this study, adult Indonesian subjects with human immunodeficiency virus (HIV) coinfected with chronic hepatitis C (CHC) will be given peginterferon alfa-2b (PEG-IFN) plus ribavirin (RBV) combination therapy. The efficacy rate (sustained virologic response, end of treatment virologic response, and sustained biochemical response), the subject morbidity rate as caused by other opportunistic infection (eg, bacterial pneumonia, tuberculosis, and other bacterial infection), and the safety and tolerability of this combination therapy will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated chronic hepatitis C with HCV-RNA positive in plasma.
* Must have finished the detoxification phase of a drug rehabilitation program and abstained for at least 6 weeks from using abused substance (alcohol, I.V. drugs and inhaled drugs) before starting therapy.
* Liver transaminases (alanine aminotransferase [ALT]) 1.5-fold above the upper limit of normal.
* Controlled HIV infection with a viral load <10,000 copies/mL and a CD4 cell (T-cell) count >200 x 10^6 cells/L, in response to a stable antiretroviral treatment (ART) or without ART if it is not required.
* Compensated liver disease with protocol-specified minimum hematologic, biochemical, and serologic criteria at the Entry visit.
* Alpha-fetoprotein value within normal limits obtained within one year prior to entry. Results above the upper limit of normal but <=50 ng/mL require both of the following: Alpha-fetoprotein value <=50 ng/mL obtained within 3 months prior to entry in the study and Ultrasound obtained within 3 months prior to entry in the study or that is negative for evidence of hepatocellular carcinoma.
* Liver biopsy (optional) within 12 months prior to study entry with a pathology report confirming that the histologic diagnosis is consistent with chronic hepatitis.
* Women of childbearing potential must be using an acceptable method of birth control or be surgically sterilized.
* Reconfirmation that sexually active males must be practicing acceptable methods of contraception during the treatment period and for 6 months after discontinuation of therapy.
* Subjects must be free of any clinically significant diseases other than hepatitis or HIV infection that would interfere with study evaluations.

Exclusion Criteria:

* Suspected hypersensitivity to interferon, PEG-interferon, or ribavirin.
* HIV therapy using didanosine (ddI) and stavudine (d4T) in their HIV medications, due to the potentiality of the resulting lactic acidosis.
* Participation in any other clinical trial within 30 days of entry to this protocol.
* Treatment with any investigational drug within 30 days of entry to this protocol.
* Subjects with organ transplants other than cornea and hair transplant.
* Any cause for the liver disease based on subject history and biopsy (where applicable) other than chronic hepatitis C, including but not limited to coinfection with hepatitis B virus (HBV); hemochromatosis (iron deposition >2+ in liver parenchyma); alpha-1 antitrypsin deficiency; Wilson's disease; autoimmune hepatitis; alcoholic liver disease; obesity-induced liver disease.
* Hemophilia or any other condition that would prevent the subject from having a liver biopsy, including anticoagulant therapy.
* Hemoglobinopathies (eg, Thalassemia)
* Evidence of advanced liver disease such as history or presence of ascites, bleeding varices, and encephalopathy.
* Any known preexisting medical condition that could interfere with the subject's participation in and completion of the protocol such as preexisting psychiatric condition, especially severe depression, or a history of severe psychiatric disorder.
* Significant cardiovascular dysfunction within the past 6 months (eg, angina, congestive heart failure, recent myocardial infarction, severe hypertension, or significant arrhythmia). Subjects with electrocardiogram (ECG) showing clinically significant abnormalities.
* Poorly controlled diabetes mellitus.
* Chronic pulmonary disease (eg, chronic obstructive pulmonary disease).
* Immunologically mediated disease.
* Any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids.
* Clinical gout.
* Clinically significant retinal abnormalities.
* Alcohol consumption of >20 gr/day.
* Women who are pregnant or nursing.
* Subjects who have not observed the designated washout periods for any of the prohibited medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG-IFN + RBV: Peginterferon alfa-2b (PEG-IFN) + Ribavirin (RBV) therapy in previously untreated chronic Hepatitis C Virus (HCV) subjects coinfected with Human Immunodeficiency Virus (HIV)
Period: Overall Study
Arm/Group | PEG-IFN + RBV
Started | 11
Completed | 0
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | PEG-IFN + RBV
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Region of Enrollment [Number; unit: participants]
  Indonesia | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Sustained Virologic Response (SVR)
Description: Treatment duration for genotype 1 participants was 48 weeks. Treatment duration for genotypes 2 & 3 participants who had baseline hepatitis c virus ribonucleic acid [HCV-RNA] <800,000 IU/mL was 24 weeks.
  SVR was defined as plasma HCV RNA level below lower level of quanitation at the end of 24 weeks follow-up (week 48 or 72).
  The study was terminated due to low enrollment. This analysis was not performed.
Time Frame: Week 48 or Week 72 (depending on duration of treatment)
Arm/Group | PEG-IFN + RBV
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants Who Achieved Virologic Response (VR)
Description: Treatment duration for genotype 1 participants was 48 weeks. Treatment duration for genotypes 2 & 3 participants who had baseline hepatitis c virus ribonucleic acid [HCV-RNA] <800,000 IU/mL was 24 weeks.
  The study was terminated due to low enrollment. This analysis was not performed.
Time Frame: 24 Weeks or 48 Weeks (depending on duration of treatment, which was either 24 or 48 weeks)
Arm/Group | PEG-IFN + RBV
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants Experiencing Opportunistic Infection
Description: The study was terminated due to low enrollment. This analysis was not performed.
Time Frame: Throughout the study (up to 72 weeks)
Arm/Group | PEG-IFN + RBV
Number analyzed (Participants) | 0

4. Primary Outcome: Number of Participants Who Achieved Sustained Biochemical Response (SBR)
Description: Treatment duration for genotype 1 participants was 48 weeks. Treatment duration for genotypes 2 & 3 participants who had baseline hepatitis c virus ribonucleic acid [HCV-RNA] <800,000 IU/mL was 24 weeks.
  SBR was defined as the presence of normal alanine aminotransferase (ALT) values at the end of 24 weeks follow-up (week 48 or 72).
  The study was terminated due to low enrollment. This analysis was not performed.
Time Frame: Week 48 or Week 72 (depending on duration of treatment, which was either 24 or 48 weeks)
Arm/Group | PEG-IFN + RBV
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Who Died
Time Frame: Throughout the study (up to 72 weeks)
Measure: Number; unit: participants
Arm/Group | PEG-IFN + RBV
Number analyzed (Participants) | 11
participants | 0

6. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: An adverse event was defined as any untoward medical occurrence in a subject administered a pharmaceutical product, biologic (at any dose), or medical device, which did not necessarily have a causal relationship with the treatment.
Time Frame: Throughout the study (up to 72 weeks)
Measure: Number; unit: participants
Arm/Group | PEG-IFN + RBV
Number analyzed (Participants) | 11
participants | 10

ADVERSE EVENTS:
Description: There was one event, "Hypertrophy Concanasalii Sinitra" that could not be coded.
Arm/Group | PEG-IFN + RBV
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN + RBV (N=11)
Anemia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN + RBV (N=11)
Anemia (Blood and lymphatic system disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Asthenopia (Eye disorders) | 1
Gastritis (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Influenza like illness (General disorders) | 7
Fatigue (General disorders) | 1
Skin infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to low enrollment. The primary and secondary outcomes were not evaluated. A formal safety analysis was not performed for the 11 participants enrolled in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator agrees not to publish/present any interim results without sponsor's prior written consent and agrees to provide sponsor 45 days written notice prior to submission for publication/presentation to permit the sponsor to review copies. The sponsor shall have the right to review and comment, including editing.